CLINICAL TRIAL: NCT04478695
Title: A Phase 1b Study Assessing Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of AMG 330 cIV in Combination With Pembrolizumab in Adult Subjects With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Study of AMG 330 in Combination With Pembrolizumab in Adult With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Amgen Decision
Sponsor: Amgen (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20170646; KEYNOTE-613 (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-06

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — AMG 330; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: AMG 330; Drug: Pembrolizumab
- Cohort 2 (Experimental)
  Interventions: Drug: AMG 330; Drug: Pembrolizumab

INTERVENTIONS:
Drug: AMG 330 — Continuous intravenous (IV) infusion.
Drug: Pembrolizumab — Intravenous (IV) infusion.

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of AMG 330, administered in combination with pembrolizumab, in participants with relapsed or refractory acute myeloid leukemia (R/R AML).

DETAILED DESCRIPTION:
This study will assess the safety and tolerability of AMG 330 in combination with pembrolizumab and whether pembrolizumab will enhance the anti-AML activity of AMG 330. Both cohort 1 and 2 will include AMG 330 and pembrolizumab with the difference being the initiation date for pembrolizumab treatment.

ELIGIBILITY:
Key Inclusion criteria

* AML as defined by the WHO Classification persisting or recurring following one or more treatment courses. Except APL
* Eastern Cooperative Oncology Group (ECOG) ≤1

Key Exclusion criteria

* Active extramedullary AML in the central nervous system.
* Known hypersensitivity to immunoglobulins.
* Non-manageable graft versus host disease.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - City of Hope National Medical Center, Duarte, California
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 participant was enrolled into this study at 1 center in the United States.
Pre-assignment Details: Screening tests and procedures were performed within the 14 days preceding administration of the first dose.
Groups:
- Cohort 1: Cohort 1 were planned to receive escalating doses of AMG 330 via continuous intravenous infusion (cIV) from Day 1 of Cycle 1 (Cycle 1 was 77 days; subsequent cycles were 57 days) for up to 6 months. The starting dose of AMG 330 was 10 μg/day, increasing up to a maximum of 600 μg/day. Cohort 1 were planned to receive 8 mg of dexamethasone 1 hour prior to each step dose of AMG 330. If the participant did not experience a dose-limiting toxicity (DLT) by Day 14, they then were also planned to receive 200 mg of pembrolizumab once every 3 weeks (Q3W) by a 30-minute intravenous (IV) infusion from Day 15 onwards. At the end of Cycle 1, there was a planned 1-week interval without administration of AMG 330, known as the infusion-free period.
- Cohort 2: Cohort 2 were planned to receive escalating doses of AMG 330 via cIV from Day 1 of Cycle 1 (cycles were 57 days) for up to 6 months. The starting dose of AMG 330 was planned to be 10 μg/day, increasing up to a maximum of 600 μg/day. The participants were also planned to receive 8 mg of dexamethasone 1 hour prior to each step dose of AMG 330, and 200 mg of pembrolizumab Q3W by a 30-minute IV infusion from Day 1 onwards. At the end of Cycle 1, there was planned to be a 1-week interval without administration of AMG 330 known as the infusion-free period..
  The trial was terminated early and 0 participants were enrolled into Cohort 2.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 1 | 0
Received AMG 330 | 1 | 0
Received Pembrolizumab | 0 | 0
Received Dexamethasone | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated with only 1 participant enrolled into Cohort 1 (0 participants were enrolled into Cohort 2). No data are reported here to maintain participant confidentiality.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male [unit: participants]
Ethnicity (NIH/OMB) [unit: participants]
Race (NIH/OMB) [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as any of the events described below occurring in a participant during the DLT window, unless clearly attributable to causes other than investigational product:
  Any treatment-related death, Grade 4 neutropenia, Grade 3-4 non hematologic toxicity not clearly resulting from the underlying leukemia, with some exceptions, cytokine release syndrome, and any Grade 5 toxicity.
Time Frame: 28 days
Population: Measured in the Dose-limiting Toxicity Evaluable Analysis Set, which was defined as DLT-evaluable participants in the Safety Analysis Set.
  The study was terminated with only 1 participant enrolled into Cohort 1 (0 participants were enrolled into Cohort 2). No data is reported here to maintain participant confidentiality.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment that occurred after first dose. Any clinically significant changes in vital signs, electrocardiograms (ECGs), and clinical laboratory tests that occurred after first dose were recorded as TEAEs.
Time Frame: From first dose of study treatment until 30 days after last dose, or end of study, whichever was earlier; median (min, max) duration was 0.79 (0.79, 0.79) months.
Population: Measured in the Safety Analysis Set, which was defined as all participants that were enrolled and received at least 1 dose of AMG 330 or pembrolizumab.
  The study was terminated with only 1 participant enrolled into Cohort 1 (0 participants were enrolled into Cohort 2). No data is reported here to maintain participant confidentiality.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Participants Who Experienced Treatment-related Adverse Events (TRAEs)
Description: A TRAE was defined as any untoward medical occurrence in a clinical study participant considered to have a possible causal relationship with the study treatment. Any clinically significant changes in vital signs, electrocardiograms (ECGs), and clinical laboratory tests that were considered to have a possible causal relationship with the study treatment were recorded as TRAEs.
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Complete Remission Without Minimal Residual Disease (CRMRD-)
Description: CRMRD- was measured according to the 2017 European Leukemia Net (ELN) criteria (Döhner et al, 2017). CRMRD- was defined as complete remission (CR) with negativity for a genetic marker by quantitative reverse transcription polymerase chain reaction (RT-qPCR), or CR with negativity by multiparametric flow cytometry (MFC). CR was defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count (ANC) ≥ 1.0 x 109/L (1000/μL); platelet count ≥ 100 x 109/L (100 000/μL).
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Complete Remission (CR)
Description: CR was measured according to the 2017 European Leukemia Net (ELN) criteria (Döhner et al, 2017). CR was defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count (ANC) ≥ 1.0 x 109/L (1000/μL); platelet count ≥ 100 x 109/L (100 000/μL).
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: CR With Incomplete Recovery (CRi)
Description: CRi was measured according to the 2017 European Leukemia Net (ELN) criteria (Döhner et al, 2017). CRi was defined as all CR criteria (bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count (ANC) ≥ 1.0 x 109/L (1000/μL); platelet count ≥ 100 x 109/L [100 000/μL]), except for residual neutropenia (< 1.0 x 109/L [1000/μL]) or thrombocytopenia (< 100 x 109/L [100 000/μL]).
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Morphological Leukemia-free State (MLFS)
Description: MLFS was measured according to the 2017 European Leukemia Net (ELN) criteria (Döhner et al, 2017). MLFS was defined as bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required.
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Partial Remission (PR)
Description: PR was measured according to the 2017 European Leukemia Net (ELN) criteria (Döhner et al, 2017). PR was defined as all hematologic criteria of CR; decrease of bone marrow blast percentage to 5 to 25%; and decrease of pre-treatment bone marrow blast percentage by at least 50%.
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Duration of Response (DoR)
Description: DoR was calculated for participants who achieved overall response (CRMRD-, CR, CRi, PR or MLFS). DoR was defined as time from the first observation indicating an objective response to the subsequent date of disease progression or death, whichever is earlier.
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Plasma Concentration of AMG 330
Time Frame: Pre-dose, 6hrs post-dose Day 1 to 71 of Cycle 1 (Cycle 1=77 days), pre-dose, 6hrs post-dose Day 1 to 50 of Cycles 2+ (Cycle 2+=57 days); end of infusion,0.5,2,4 and 8hrs post-infusion on Days 78 and 57 of Cycle 1 and 2 infusion-free periods respectively
Population: Measured in the Pharmacokinetic (PK) Analysis Set which contained all participants who received at least 1 dose of AMG 330 or pembrolizumab and had at least 1 PK sample collected.
  The study was terminated with only 1 participant enrolled into Cohort 1 (0 participants were enrolled into Cohort 2). No data is reported here to maintain participant confidentiality.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Half-life of AMG 330
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Steady State Concentration of AMG 330
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Volume of Distribution of AMG 330
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Clearance of AMG 330
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants With Anti-AMG 330 Antibody Formation
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Mortality reporting was from enrollment until end of study; median (min, max) duration was 0.82 (0.82, 0.82) months.
Description: All-cause mortality is reported for all enrolled participants. The study was terminated with only 1 participant enrolled into Cohort 1 (0 participants were enrolled into Cohort 2). No serious adverse event or other adverse event data is reported here to maintain participant confidentiality.
Arm/Group | Cohort 1
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This study was early terminated, leading to a small number of participants enrolled and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT04478695/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT04478695/SAP_001.pdf